CLINICAL TRIAL: NCT02139969
Title: GreenLight XPS Laser System for the Treatment of Benign Prostatic Hyperplasia: Evaluation of Safety, Efficacy, and Quality of Life Through Retrospective Chart Review
Brief Title: GreenLight XPS Laser System Retrospective Chart Review
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: PE1401
Record Dates: First submitted 2014-05-13; First posted 2014-05-16 (Estimated); Results first posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2018-01

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- GreenLight XPS Laser System: Treatment of BPH in men using the GreenLight XPS Laser System and the MoXy fiber
  Interventions: Device: GreenLight XPS Laser System

INTERVENTIONS:
Device: GreenLight XPS Laser System

SUMMARY:
The purpose of this study is to gain information on the safety, efficacy, and quality of life in subjects who have had the GreenLight XPS procedure.

DETAILED DESCRIPTION:
This is a retrospective chart review conducted at six centers in the United States and Canada. This review will evaluate the safety and efficacy of GreenLight XPS in subjects who received treatment on or after 01-Aug-2010.

ELIGIBILITY:
Inclusion Criteria:

* Men who have had a GreenLight XPS procedure with a MoXy Fiber since 01-Aug-2010.

Exclusion Criteria:

* Subject has had prior radiation.
* Subject has a diagnosis of neurogenic bladder confirmed by urodynamic studies (BOO, detrusor overactivity (DO), impaired detrusor contractor (IDC))
* Subject has a neurologic disorder that would impact bladder function (MS, Parkinson, Spinal Cord Injury) (note: Stroke patients not excluded)
* Subject has an artificial urinary sphincter

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of males who have had the GreenLight XPS procedure with the MoXy fiber on or after 01-Aug-2010. The cohort will be selected from six pre-selected urology clinics in the US and one pre-selected urology clinic in Canada.
Sampling Method: Non-Probability Sample
Enrollment: 956 (Actual)
Dates: Start 2014-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mahmood A. Hai, M.D., Principal Investigator — Affiliates Division, Comprehensive Urology
Locations (6):
- United States (5):
  - El Camino Urology Medical Group, Inc., Mountain View, California
  - Georgia Urology, Atlanta, Georgia
  - Affiliates Division, Comprehensive Urology, Westland, Michigan
  - Houston Metro Urology, Houston, Texas
  - Urology of Virginia, PLLC, Virginia Beach, Virginia
- University of Montreal Hospital Center, Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- GreenLight XPS Laser System: Treatment of men with BPH using the GreenLight XPS Laser System and the MoXy fiber
Period: Overall Study
Arm/Group | GreenLight XPS Laser System
Started | 956
Completed | 956
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- GreenLight XPS Laser System: Treatment of BPH in men using the GreenLight XPS Laser System
Arm/Group | GreenLight XPS Laser System
Number analyzed (Participants) | 956
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.6 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 956
Region of Enrollment [Number; unit: participants]
  Canada | 199
  United States | 757

OUTCOME MEASURES:

1. Primary Outcome: International Prostate Symptom Score (IPSS)
Description: Evaluate the proportion of subjects who have mild or no BPH symptoms at six months post-procedure; e.g. an IPSS of eight or less at 6-month follow-up. An IPSS of eight or less indicates the subject is asymptomatic or has mild symptoms, a score of 9-21 indicates the subject has moderate symptoms, and a score of >21 indicates the subject has severe symptoms. IPSS scores can range from 0-35.
Time Frame: 6 months post-procedure
Population: This study was retrospective chart review of available data collected in the medical records. The intention was to collect and analyze data through five years post-procedure; however, the data collected was minimal. Results posted here are reflective of the results that have been published (through 6-months).
Measure: Count of Participants; unit: Participants
Arm/Group | GreenLight XPS Laser System
Number analyzed (Participants) | 572
Participants
  Score of <=8 | 437
  Score of 9-21 | 118
  Score of >21 | 17

2. Primary Outcome: Occurrence of Adverse Events Related to the Study Treatment.
Description: Treatment-related adverse events include:
  * Event related to the study device or procedure
  * Intra-operative adverse event related to the study device or procedure
  * Serious adverse events related to the study device or procedure
  The number of events as well as the number and percentage of subjects with the event will be calculated.
Time Frame: 365 Days
Population: Number of participants with a treatment-related adverse event.
Measure: Number; unit: Treatment-related Events
Arm/Group | GreenLight XPS Laser System
Number analyzed (Participants) | 191
Treatment-related Events | 249

3. Secondary Outcome: Characteristics of the Study Procedure
Description: Summary of the study procedure, including length of procedure and lasing time
Time Frame: Participants will be followed from admission through discharge from the medical facility, an expected average of 2 days.
Population: Data collected for this study was retrospective in nature and only data available in the medical records could be reported.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | GreenLight XPS Laser System
Number analyzed (Participants) | 956
minutes
  Length of Procedure (minutes): number analyzed (Participants) | 906
  Length of Procedure (minutes) | 57.1 (28.6)
  Lasing Time (minutes): number analyzed (Participants) | 952
  Lasing Time (minutes) | 33.2 (18.9)

4. Secondary Outcome: Characteristics of the Study Procedure and Immediate Outcomes
Description: Summary of characteristics of the study procedure and immediate outcomes: total energy used (kJ)
Time Frame: Participants will be followed from admission through discharge from the medical facility, an expected average of 2 days.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kJ
Arm/Group | GreenLight XPS Laser System
Number analyzed (Participants) | 954
kJ | 275.8 (180.7)

5. Secondary Outcome: Assess Changes in Quality of Life Related to BPH Symptoms.
Description: Summarize IPSS-QOL from baseline through six months post-procedure for all data available during the retrospective review. The quality of life assessment responses includes: Delighted, Pleased, Mostly Satisfied, Mixed-neither satisfied or dissatisfied, Mostly Dissatisfied, Unhappy, or Terrible (range of 0 to 6).The results presented below represent the change from baseline to six months post-procedure for any response. Lower scores indicate a better outcome.
Time Frame: Baseline through six months post-procedure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GreenLight XPS Laser System
Number analyzed (Participants) | 956
units on a scale | 1.3 (1.3)

6. Secondary Outcome: Assess Changes in Objective Measures of Urologic Function.
Description: Changes in objective measures of urologic function from baseline through six months post-procedure using Peak Flow Rate (Qmax)
Time Frame: Baseline through six months post-procedure.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ml/sec
Arm/Group | GreenLight XPS Laser System
Number analyzed (Participants) | 956
ml/sec
  Peak Flow Rate (Qmax) Baseline (ml/sec): number analyzed (Participants) | 707
  Peak Flow Rate (Qmax) Baseline (ml/sec) | 8.7 (5.7)
  Qmax 6 months (ml/sec): number analyzed (Participants) | 409
  Qmax 6 months (ml/sec) | 18.0 (8.9)
  Qmax Change from Baseline: number analyzed (Participants) | 354
  Qmax Change from Baseline | 10.9 (10.0)

7. Secondary Outcome: Number of Participants With ER Visits, Hospital Admissions, and Surgical Re-treatments for Treatment-related Adverse Events Up to 90 Days Post-Procedure
Description: * Emergency room visit for an adverse event related to the study device or procedure within 90 days of procedure
  * Hospital admission for an adverse event related to the study device or procedure within 90 days of procedure
  * Surgical intervention for an adverse event related to the study device or procedure within 90 days of procedure
Time Frame: Up to 90 days post-procedure.
Population: Data collected for this study was retrospective in nature and only data available in the medical records could be reported. Results presented are number of subjects.
Measure: Number; unit: Participants
Arm/Group | GreenLight XPS Laser System
Number analyzed (Participants) | 956
Participants
  ER Visit 30 Days | 39
  ER Visit 90 Days | 43
  Hospital Admission 30 Days | 14
  Hospital Admission 90 Days | 19
  Surgical Re-treatment 90 Days | 4

8. Secondary Outcome: Evaluate the Percentage of Participants Experience Ongoing Treatment-related Urinary Incontinence
Description: The percentage (count/n) of subjects with an ongoing urinary incontinence event at 90 and 180 days post-procedure. An incontinence event is considered ongoing if the onset was on or before the specified time point and the event is either unresolved or resolved after that time point.
Time Frame: 90 days, 180 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of incontinence events
Arm/Group | GreenLight XPS Laser System
Number analyzed (Participants) | 956
percentage of incontinence events
  Incontinence, Stress 90 Days: number analyzed (Participants) | 898
  Incontinence, Stress 90 Days | 0.9 [0.4 to 1.7]
  Incontinence, Urge 90 Days: number analyzed (Participants) | 898
  Incontinence, Urge 90 Days | 0.9 [0.4 to 1.7]
  Incontinence, Stress 180 Days: number analyzed (Participants) | 850
  Incontinence, Stress 180 Days | 1.3 [0.6 to 2.3]
  Incontinence, Urge 180 Days: number analyzed (Participants) | 851
  Incontinence, Urge 180 Days | 1.1 [0.5 to 2.0]

9. Secondary Outcome: Assess the Occurrence of Surgical Retreatment for BPH in GreenLight XPS Patients.
Description: Number of surgical re-treatment for BPH as a result of prostate tissue regrowth or insufficient prostatic tissue removal.
Time Frame: Procedure through five years post-procedure.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GreenLight XPS Laser System
Number analyzed (Participants) | 955
Participants
  Reobstruction due to prostate regrowth | 4
  Insufficient tissue removal | 3

10. Secondary Outcome: Characteristics of the Study Procedure and Immediate Outcomes
Description: Summarize characteristics of the study procedure and immediate outcomes: length of catheterization
Time Frame: Participants will be followed from admission through discharge from the medical facility, an expected average of 2 days.
Population: as for outcome 3
Measure: Mean (Full Range); unit: days
Arm/Group | GreenLight XPS Laser System
Number analyzed (Participants) | 709
days | 1.2 [0.1 to 14.0]

11. Secondary Outcome: Length of Hospital Stay
Description: Summarize length of hospital stay (in days) from admission through discharge
Time Frame: The number of days from admission through discharge from the medical facility will be measured.
Population: as for outcome 3
Measure: Mean (Full Range); unit: days
Arm/Group | GreenLight XPS Laser System
Number analyzed (Participants) | 817
days | 0.5 [0.1 to 6.1]

12. Secondary Outcome: Type of Hospital Stay
Description: Summarize characteristics of the type of hospital stay (in-patient vs out-patient with an overnight stay)
Time Frame: Data will be collected during the time of their hospital stay from admission through discharge
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | GreenLight XPS Laser System
Number analyzed (Participants) | 954
participants
  Admission Type: Outpatient | 674
  Admission Type: Outpatient overnight stay | 222
  Admission Type: inpatient | 58

13. Secondary Outcome: Number of Participants Stratified by Number of Fibers Used During Procedure
Description: Summarize characteristics of the study procedure and immediate outcomes: number of fibers used
Time Frame: Participants will be followed from admission through discharge from the medical facility, an expected average of 2 days.
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | GreenLight XPS Laser System
Number analyzed (Participants) | 953
participants
  Number of Fibers Used: 1 | 873
  Number of Fibers Used: 2 | 76
  Number of Fibers Used: >=3 | 4

14. Secondary Outcome: Assess Changes in Objective Measures of Urologic Function
Description: Changes in objective measures of urologic function from baseline through six months post-procedure using post void residual
Time Frame: Baseline through six months post-procedure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | GreenLight XPS Laser System
Number analyzed (Participants) | 956
ml
  PVR Baseline (ml): number analyzed (Participants) | 811
  PVR Baseline (ml) | 204.3 (221.2)
  PVR 6 Months (ml): number analyzed (Participants) | 583
  PVR 6 Months (ml) | 46.1 (95.2)
  PVR Change from Baseline: number analyzed (Participants) | 511
  PVR Change from Baseline | -172 (215.4)

15. Secondary Outcome: Changes in Objective Measures of Urologic Function
Description: Changes in objective measures of urologic function from baseline through six months post-procedure using prostate volume
Time Frame: Baseline through six months post-procedure.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | GreenLight XPS Laser System
Number analyzed (Participants) | 956
grams
  Prostate Volume (g) Baseline: number analyzed (Participants) | 804
  Prostate Volume (g) Baseline | 76.0 (49.0)
  Prostate Volume (g) 6 Months: number analyzed (Participants) | 148
  Prostate Volume (g) 6 Months | 44.0 (36.2)
  Prostate Volume (g) Change from Baseline: number analyzed (Participants) | 141
  Prostate Volume (g) Change from Baseline | -31.8 (38.3)

16. Secondary Outcome: Assess Changes in Objective Measures of Urologic Function.
Description: Changes in objective measures of urologic function from baseline through six months post-procedure using prostate specific antigen
Time Frame: From baseline through six months post-procedure.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | GreenLight XPS Laser System
Number analyzed (Participants) | 956
ng/ml
  PSA (ng/ml) Baseline: number analyzed (Participants) | 639
  PSA (ng/ml) Baseline | 4.9 (7.8)
  PSA (ng/ml) 6 Months: number analyzed (Participants) | 499
  PSA (ng/ml) 6 Months | 2.6 (7.6)
  PSA (ng/ml) Change from Baseline: number analyzed (Participants) | 394
  PSA (ng/ml) Change from Baseline | -2.0 (7.1)

ADVERSE EVENTS:
Time Frame: Any device or treatment related adverse event was collected during the retrospective chart review, up to five years post-procedure for each participant.
Arm/Group | GreenLight XPS Laser System
Serious Adverse Events (participants affected / at risk) | 13/956
Other Adverse Events (participants affected / at risk) | 182/956
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GreenLight XPS Laser System (N=956)
Intraoperative Bleeding (Renal and urinary disorders) | 1 (1)
Bladder Neck Obstruction (Renal and urinary disorders) | 4 (4)
Hematuria - Gross (Renal and urinary disorders) | 2 (2)
Irritative Voiding Symptoms (Renal and urinary disorders) | 2 (2)
Urinary Retention (Renal and urinary disorders) | 2 (2)
Clot Retention (Renal and urinary disorders) | 1 (1)
Reobstruction Due to Prostate Regrowth (Renal and urinary disorders) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
Other (General disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GreenLight XPS Laser System (N=956)
Urinary Incontinence - De Novo Stress (Renal and urinary disorders) | 13 (13)
Urinary Incontinence - De Novo Urge (Renal and urinary disorders) | 13 (13)
Urinary Tract Infection (Renal and urinary disorders) | 29 (29)
Erectile Dysfunction - De Novo (Renal and urinary disorders) | 1 (1)
Bladder Neck Obstruction (Renal and urinary disorders) | 10 (10)
Dysuria (Renal and urinary disorders) | 16 (16)
Irritative Voiding Symptoms (Renal and urinary disorders) | 13 (13)
Urinary Frequency (Renal and urinary disorders) | 9 (9)
Urinary Retention (Renal and urinary disorders) | 39 (39)
Urinary Urgency (Renal and urinary disorders) | 19 (19)
Bladder Injury (Renal and urinary disorders) | 1 (1)
Urethral Injury (Renal and urinary disorders) | 2 (2)
Urinary Incontinence - Worsening Urge (Renal and urinary disorders) | 1 (1)
Erectile Dysfunction - Worsening (Renal and urinary disorders) | 1 (1)
Bladder Spasms (Renal and urinary disorders) | 1 (1)
Hematospermia (Renal and urinary disorders) | 1 (1)
Hematuria - Gross (Renal and urinary disorders) | 8 (8)
Prostatitis (Renal and urinary disorders) | 1 (1)
Nocturia (Renal and urinary disorders) | 1 (1)
Clot Retention (Renal and urinary disorders) | 9 (9)
Fever (General disorders) | 1 (1)
Cardiac Arrhthmia (Cardiac disorders) | 2 (2)
Other (General disorders) | 1 (1)
Retrograde Ejaculation - De Novo (Renal and urinary disorders) | 18 (18)
Urethral Stricture (Renal and urinary disorders) | 6 (6)
Insufficient Tissue Removal (Renal and urinary disorders) | 3 (3)
Malfunction of XPS Fiber (Renal and urinary disorders) | 3 (3)
Reobstruction Due to Prostate Regrowth (Renal and urinary disorders) | 3 (3)
Excessive Bleeding (Renal and urinary disorders) | 2 (2)
Intraoperative Bleeding (Renal and urinary disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 1 (1)
Perforation - Prostate (Renal and urinary disorders) | 1 (1)
Renal Failure / Insufficiency (Renal and urinary disorders) | 1 (1)
Sloughing (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No